CLINICAL TRIAL: NCT04115514
Title: PHASE II RANDOMIZED, INTERVENTION VERSUS NON- INTERVENTION, MULTI- CENTER STUDY OF THE EFFECTS OF THYROID HORMONE (T3) ON SAFETY/TOLERABILITY AND OXYGENATION IN SUBJECTS WITH ACUTE RESPIRATORY DISTRESS SYNDROME (ARDS)
Brief Title: Treatment of ARDS With Instilled T3
Acronym: ARDS+T3
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PACS-2020-23242
Record Dates: First submitted 2019-03-12; First posted 2019-10-04 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: ARDS, Human; Lung, Wet; Thyroid; Pulmonary Edema; Lung Inflammation
MeSH Terms: conditions — Respiratory Distress Syndrome; Pulmonary Edema; Thyroid Diseases; Pneumonia | interventions — Triiodothyronine

STUDY DESIGN:
Intervention Model Description: Randomized, unblinded, intervention versus non-intervention trial. 68 [50 treatment + 18 controls]
Masking Description: None applicable
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Experimental): Liothyronine Sodium (T3+0.9% sodium chloride) modified formulation specifically for airway instillation.
  Interventions: Drug: Liothyronine Sodium (T3+0.9% sodium chloride) modified formulation specifically for airway instillation.
- Control arm (Other): Standard of Care
  Interventions: Other: Non-intervention

INTERVENTIONS:
Drug: Liothyronine Sodium (T3+0.9% sodium chloride) modified formulation specifically for airway instillation. — Study Drug Administration:
  * Dose/Volume- Liothyronine Sodium 50 mcg / 10 mL
  * Frequency/Duration: Twice daily over 5 days (10 total doses), or until extubation, whichever comes first.
  * Method: Instilled via a catheter through the ETT directly into the airway.
  Arms: Treatment Arm
Other: Non-intervention — Standard of Care (SOC)
  Arms: Control arm

SUMMARY:
It is hypothesized that instillation of Liothyronine Sodium (T3) into the airspace will be safe, well tolerated, and will increase alveolar fluid clearance and decrease inflammation in patients with ARDS, reflected in improved oxygenation index (OI) and oxygenation saturation index (OSI).

DETAILED DESCRIPTION:
T3 Therapy in ARDS- Phase 2 Randomized, Unblinded, Intervention versus Non- Intervention Trial. Enrollment 68 participants (50 treatment + 18 control). Purpose- To determine the safety and tolerability of T3 delivery into the lungs of ARDS patients, and to measure the effect of T3 on Oxygenation in ARDS patients. Study Drug- Liothyronine Sodium (T3), 50 mcg will be instilled twice daily via a catheter through the ETT into the airway in a total volume of 10 mL (T3+0.9% sodium chloride), over 5 days (10 total doses), or until extubation, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

Study population is critically ill patients requiring mechanical ventilatory support for ARDS in an intensive care unit.

* Adults (≥18 years of age).
* Male or female (non-pregnant).
* Clinical diagnosis of ARDS (all are required):

  1. Onset: <= 7 days.
  2. Chest x-ray: Bilateral Patchy Opacities, Infiltrates.
  3. Mechanical Vent Support: PEEP or CPAP Support >= 5 cm H2O.
  4. Pulmonary Edema: Not fully explained by cardiogenic etiology.
  5. Hypoxia: PaO2/FIO2 Ratio <300, or O2Sat/FIO2 Ratio <315.
* On mechanical ventilatory support.
* Capable of giving informed consent directly or from the subject's legally authorized representative (LAR) as determined by the site Principal Investigator and/or Sub- Investigators.

Exclusion Criteria:

Patients with any of the following conditions will be excluded from this trial:

* Inadequate medical history for determining inclusion/exclusion criteria, as determined by the Principal Investigator and/or Sub- Investigators.
* Unlikely to complete the protocol with clinic follow-up after discharge, as determined by the Principal Investigator and/or Sub- Investigators or hospice status.
* Prior history of thyroid cancer or hyperthyroidism, per thorough patient/family interviews, review of past medical history, medication list, laboratory test.
* Prior history of cardiovascular disease defined as:

  1. Hypertensive crisis in the past 3 months (systolic >200, or diastolic >120 mmHg),
  2. Sustained ventricular arrhythmia in the past 3 months (duration >30 seconds)
  3. Coronary artery disease (documented >=70% occlusion untreated in any coronary vessel), as per the 2021 ACC/AHA/SCAI Guidelines for Coronary Artery Revascularization.
  4. Cardiac-related angina pectoris (>=2 episodes in the past 3 months)
  5. Myocardial infarction with ischemia on ECG (i.e.,new ST- elevation/depression of >1mm in contiguous leads).
  6. Peripheral vascular disease (documented >=70% occlusion untreated in any peripheral vessel), as per the 2018 ACC/AHA/SCAI/SIR/SVM Guidelines for Appropriate Use Criteria for Peripheral Artery Intervention.
  7. Decompensated or symptomatic heart failure (i.e., hospitalized for CHF exacerbation, or a change in CHF medications within two weeks prior)
* Currently pregnant or breastfeeding.
* Known allergy to study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2020-03-30 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Oxygenation: Oxygenation Index (OI), and/or Oxygenation Saturation Index (OSI). | baseline
  To assess the efficacy of airway instilled T3 improving oxygenation by reducing OI and OSI in ARDS patients. OI will be measured by mechanical ventilator (FIO2 and Mean Airway Pressure, MAP), and ABG (PaO2). OSI will be measured by mechanical ventilator (FIO2, SpO2 and MAP):
  OI = (FIO2 x MAP / PaO2). OSI = (FIO2 x MAP / SpO2).
Oxygenation: Oxygenation Index (OI), and/or Oxygenation Saturation Index (OSI). | 6 hours post-dose
  To assess the efficacy of airway instilled T3 improving oxygenation by reducing OI and OSI in ARDS patients. OI will be measured by mechanical ventilator (FIO2 and Mean Airway Pressure, MAP), and ABG (PaO2). OSI will be measured by mechanical ventilator (FIO2, SpO2 and MAP):
  OI = (FIO2 x MAP / PaO2). OSI = (FIO2 x MAP / SpO2).
Oxygenation: Oxygenation Index (OI), and/or Oxygenation Saturation Index (OSI). | 12 hours post-dose
  To assess the efficacy of airway instilled T3 improving oxygenation by reducing OI and OSI in ARDS patients. OI will be measured by mechanical ventilator (FIO2 and Mean Airway Pressure, MAP), and ABG (PaO2). OSI will be measured by mechanical ventilator (FIO2, SpO2 and MAP):
  OI = (FIO2 x MAP / PaO2). OSI = (FIO2 x MAP / SpO2).
Oxygenation: Oxygenation Index (OI), and/or Oxygenation Saturation Index (OSI). | 24 hours post-dose
  To assess the efficacy of airway instilled T3 improving oxygenation by reducing OI and OSI in ARDS patients. OI will be measured by mechanical ventilator (FIO2 and Mean Airway Pressure, MAP), and ABG (PaO2). OSI will be measured by mechanical ventilator (FIO2, SpO2 and MAP):
  OI = (FIO2 x MAP / PaO2). OSI = (FIO2 x MAP / SpO2).
Oxygenation: Oxygenation Index (OI), and/or Oxygenation Saturation Index (OSI). | 48 hours post-dose
  To assess the efficacy of airway instilled T3 improving oxygenation by reducing OI and OSI in ARDS patients. OI will be measured by mechanical ventilator (FIO2 and Mean Airway Pressure, MAP), and ABG (PaO2). OSI will be measured by mechanical ventilator (FIO2, SpO2 and MAP):
  OI = (FIO2 x MAP / PaO2). OSI = (FIO2 x MAP / SpO2).
Oxygenation: Oxygenation Index (OI), and/or Oxygenation Saturation Index (OSI). | 72 hours post-dose
  To assess the efficacy of airway instilled T3 improving oxygenation by reducing OI and OSI in ARDS patients. OI will be measured by mechanical ventilator (FIO2 and Mean Airway Pressure, MAP), and ABG (PaO2). OSI will be measured by mechanical ventilator (FIO2, SpO2 and MAP):
  OI = (FIO2 x MAP / PaO2). OSI = (FIO2 x MAP / SpO2).
Oxygenation: Oxygenation Index (OI), and/or Oxygenation Saturation Index (OSI). | 96 hours post-dose
  To assess the efficacy of airway instilled T3 improving oxygenation by reducing OI and OSI in ARDS patients. OI will be measured by mechanical ventilator (FIO2 and Mean Airway Pressure, MAP), and ABG (PaO2). OSI will be measured by mechanical ventilator (FIO2, SpO2 and MAP):
  OI = (FIO2 x MAP / PaO2). OSI = (FIO2 x MAP / SpO2).
Oxygenation: Oxygenation Index (OI), and/or Oxygenation Saturation Index (OSI). | 120 hours post-dose
  To assess the efficacy of airway instilled T3 improving oxygenation by reducing OI and OSI in ARDS patients. OI will be measured by mechanical ventilator (FIO2 and Mean Airway Pressure, MAP), and ABG (PaO2). OSI will be measured by mechanical ventilator (FIO2, SpO2 and MAP):
  OI = (FIO2 x MAP / PaO2). OSI = (FIO2 x MAP / SpO2).

SECONDARY OUTCOMES:
Pulmonary events | baseline and 120 hours post-dose
  Progressive hemoptysis: bright, red blood in streaks, mixed or clots within sputum on suctioning of greater than 30 mL accumulation anytime following the initial and subsequent intratracheal dosing administrations.
Cardiovascular event 1 | baseline to 120hours post-dose
  New sustained ventricular arrhythmia (>30 secs)
Cardiovascular event 2 | baseline to 120hours post-dose
  New sustained accelerated junctional arrhythmia (rate >80 bpm) with worsened hypotension (decrease in mean arterial pressure to less than 65mmHg).
Cardiovascular event 3 | baseline to 120hours post-dose
  New sustained atrial fibrillation with rapid ventricular response (ventricular rate >160 bpm) with worsened hypotension (decrease in mean arterial pressure to less than 65mmHg).
Cardiovascular event 4 | baseline to 120hours post-dose
  Cardiac arrest (pulseless electrical activity, or asystole).
Cardiovascular event 5 | baseline to 120hours post-dose
  Hypertensive crisis (systolic pressure of 180 mmHg (or higher), or diastolic pressure of 120 mmHg (or higher) or change in MAP > 20 mmHg with three consecutive measurements over 30 minutes).
SOC pulmonary vasodilator | baseline and 5 days
  yes or no
SOC pressor(s) dose(s) | baseline and 5 days
SOC diurectic(s) dose(s) | baseline and 5 days
Ventilator Free Days | baseline and 5 days
ICU Free Days | baseline and 5 days
Oxygen Free Days | baseline and 5 days
All-Cause Mortality | baseline and 5 days
Tracheostomy placement requirement | baseline and 5 days
Supplemental oxygen on discharge | baseline and 5 days
  yes or no
Discharge disposition | baseline and 5 days
  home, inpatient rehabilitation, long-term acute care hospital (LTACH)
TSH, Total T3, Free T3, Free T4 | baseline and 156-hrs post-dose
Free T3, Free T4 | baseline and 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Timothy P Rich, MD, Study Director — University of Minnesota; David H Ingbar, MD, Study Chair — University of Minnesota; Ronald A Reikoff, MD, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - M Health Fairview Southdale Hospital, Edina, Minnesota
  - East Bank Hospital - M Health Fairview University of Minnesota Medical Center, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Flory CM, Norris BJ, Larson NA, Coicou LG, Koniar BL, Mysz MA, Rich TP, Ingbar DH, Schumacher RJ. A Preclinical Safety Study of Thyroid Hormone Instilled into the Lungs of Healthy Rats-an Investigational Therapy for ARDS. J Pharmacol Exp Ther. 2021 Jan;376(1):74-83. doi: 10.1124/jpet.120.000060. Epub 2020 Oct 30. PMID 33127750